CLINICAL TRIAL: NCT03224871
Title: UCDCC#269: A Pilot Study of Interlesional IL-2 and Hypofractionated Radiotherapy in Patients With Metastatic Non-small Cell Lung Cancer Who Are Refractory to PD 1 / PD L1 Blockade.
Brief Title: UCDCC#269: A Pilot Study of Interlesional IL-2 and RT in Patients With NSCLC.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Arta Monjazeb, Principal Investigator, University of California, Davis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1032095; UCDCC#269 (Other: UC Davis)
Record Dates: First submitted 2017-07-05; First posted 2017-07-21 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: METASTATIC NON-SMALL CELL LUNG CANCER
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aldesleukin; Interleukin-2; Nivolumab; pembrolizumab; Radiotherapy

STUDY DESIGN:
Intervention Model Description: All patients will go through the same process except that some patients will be on nivolumab as checkpoint blockade and some patients will be on pembrolizumab as checkpoint blockade.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): Intralesional IL-2, Radiotherapy will be given to all patients. Immune checkpoint blockade with Nivolumab will be started on week 1 day 1, concurrent with radiotherapy and continue with cycles every 2 weeks.
  Interventions: Drug: Intralesional IL-2; Drug: Nivolumab; Radiation: Radiotherapy
- Pembrolizumab (Experimental): Intralesional IL-2, Radiotherapy will be given to all patients. Immune checkpoint blockade with Pembrolizumab will be started on week 1 day 1, concurrent with radiotherapy and continue with cycles every 3 weeks.
  Interventions: Drug: Intralesional IL-2; Drug: Pembrolizumab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Intralesional IL-2 — High dose IL-2 (HD-IL-2) is a cytokine produced endogenously by activated T cells and is effective in the treatment of a variety of malignancies because it has both immune-modulating and antitumor properties. In an attempt to take advantage of the robust immune activating effects of IL-2 but avoid the toxicity of high dose systemic IL-2 we and others have investigated the use of intralesional IL-2 injections.
  Other Names: Proleukin; Aldesleukin; IL-2
Drug: Nivolumab — Nivolumab is a fully humanized IgG4 PD-1 blocking antibody which has shown promising efficacy as an immune checkpoint inhibitor in lung cancer. Immune checkpoint blockade will be started on week 1 day 1, concurrent with radiotherapy and continue with cycles every 2 weeks for patients on Nivolumab.
  Other Names: Opdivo
  Arms: Nivolumab
Drug: Pembrolizumab — PD-1 inhibitor. Immune checkpoint blockade will be started on week 1 day 1, concurrent with radiotherapy and continue with cycles every 3 weeks for patients on Pembrolizumab.
  Other Names: Keytruda
  Arms: Pembrolizumab
Radiation: Radiotherapy — Radiotherapy will be delivered to the treatment lesion during the first week of therapy using an 8 Gy x 3 fractions palliative regimen. Fractions may be delivered on consecutive or every other day but must be completed during week 1 and will not be repeated in future cycles.
  Other Names: Ionizing radiation therapy; Radiation therapy

SUMMARY:
The advent of checkpoint blockade immunotherapy has revolutionized the management of metastatic non-small cell lung cancer (NSCLC). Despite the promising evidence for deep and durable responses with these agents the majority of patients fail to respond. The investigators hypothesize that a novel strategy combining radiotherapy and intralesional interleukin-2 (IL-2), a signaling molecule and member of the cytokine family involved in the activation of leukocytes and lymphocytes, may overcome resistance to checkpoint blockade therapy and offer significant clinical benefit to patients who fail to respond to checkpoint blockade alone. The investigators propose a microtrial testing the feasibility of a bold combinatorial immunotherapy strategy consisting of radiotherapy (RT), intralesional IL-2, and check-point blockade for metastatic non-small cell lung cancer patients who have progressed after checkpoint inhibition. IL-2 can upregulate PD-1 expression and activate T-cells.

DETAILED DESCRIPTION:
The advent of checkpoint blockade immunotherapy has revolutionized the management of metastatic non-small cell lung cancer (NSCLC). Despite the promising evidence for deep and durable responses with these agents the majority of patients fail to respond. The investigators hypothesize that a novel strategy combining radiotherapy and intralesional interleukin-2 (IL-2), a signaling molecule and member of the cytokine family involved in the activation of leukocytes and lymphocytes, may overcome resistance to checkpoint blockade therapy and offer significant clinical benefit to patients who fail to respond to checkpoint blockade alone. The investigators propose a microtrial testing the feasibility of a bold combinatorial immunotherapy strategy consisting of radiotherapy (RT), intralesional IL-2, and check-point blockade for metastatic non-small cell lung cancer patients who have progressed after checkpoint inhibition. IL-2 can upregulate PD-1 expression and activate T-cells. There is data supporting combination therapies with IL-2 and checkpoint blockade, IL-2 and radiotherapy, and checkpoint blockade and radiotherapy but clinical data is limited and the triple combination has never been tested. IL-2 + checkpoint blockade was recently tested in a small clinical trial and showed promising results but RT was not included in this trial. As outlined above RT has been demonstrated to increase the efficacy of both IL-2 and checkpoint blockade. The investigators believe that the triple combination of radiotherapy + IL-2 + checkpoint inhibition will be highly effective as RT + IL-2 can serve highly activate the immune system and checkpoint blockade can reverse the immune suppressive pathways induced by tumor and therapy. The investigators hypothesize that the combination of intralesional IL-2 with radiotherapy will act as an "in-situ" vaccine inducing an anti-tumor immune response. The investigators further hypothesize that this vaccine effect will convert patients with primary or secondary resistance to checkpoint blockade into responders since one mechanism of resistance to checkpoint blockade appears to be lack of a pre-existing anti-tumor immune response. The primary endpoint is tolerability, safety and toxicity. Exploratory endpoints include abscopal response rate, objective response rate, disease control rate, progression free survival, and correlative studies. This trial will incorporate robust correlative assays to provide insights into mechanisms of resistance to checkpoint blockade and how this therapy may overcome that resistance. This trial, although small, has the potential to drastically advance both our understanding and treatment of metastatic lung cancer.

This is a pilot phase I study that will evaluate the safety and toxicity of this combinatorial approach. Eligible patients with NSCLC who fail to respond to PD1/PDL1 checkpoint blockade will be enrolled. Patients will continue on checkpoint blockade and receive intralesional IL-2 in combination with hypofractionated radiotherapy. Radiotherapy will be delivered to the treatment lesion during the first week of therapy using an 8 Gy x 3 fractions palliative regimen. Fractions may be delivered on consecutive or every other day but must be completed during week 1 and will not be repeated in future cycles. Immune checkpoint blockade will be started on week 1 day 1, concurrent with radiotherapy and continue with cycles every 2 (nivolumab) or 3 (pembrolizumab) weeks. A total of four Interleukin-2 treatments will be delivered into the treatment lesion by intralesional injections twice weekly starting 24-72 hours after the completion of radiotherapy and to be completed no later than study Day 21. Intralesional injections will be performed by palpation of the lesion or under ultrasound or CT guidance as indicated. Intralesional IL-2 injections will follow guidelines, which we have previously published. Briefly, each patient will receive an initial test dose of 3 x 106 IU of IL-2, which will be escalated to 7 x 106 for the second treatment and then 15 x 106 IU for the final two treatments as tolerated. If a dose level is not tolerated the treatment will be de-escalated to previous dose levels for subsequent treatments. If 3 million IU IL-2 is not tolerated the dose can be de-escalated to 1 million IU IL-2. If 1 million IU IL-2 is not tolerated the treatment will be deemed intolerable and patient removed from study.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age with histologically proven NSCLC.
2. Failure to respond to standard of care checkpoint blockade therapy or previously responding patients who progress on checkpoint blockade therapy.
3. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 - 2 (Appendix 1)
4. Presence of a candidate treatment lesion (subcutaneous or nodal lesions are preferable but visceral lesions will be considered) accessible and safe for radiotherapy and serial intralesional injections.
5. Presence of at least one target lesion (distinct from treatment lesion and outside of treatment lesion radiation field) evaluable for response by RECIST 1.1
6. Life expectancy ≥ 6 months
7. The following laboratory results obtained within 14 days of the first study treatment:

   * ANC > 1500 cells/ul
   * WBC count > 2500/uL
   * Lymphocyte count >500/uL
   * Platelet count > 100,000/uL
   * Hemoglobin > 9 g/dL
8. Liver function tests meeting one of the following criteria:

   * AST and ALT < 2.5 x ULN with alkaline phosphatase < 2.5 x ULN OR
   * AST and ALT < 1.5 x ULN, with alkaline phosphatase > 2.5 x ULN
9. Serum bilirubin ≤ 1.0 x ULN.
10. INR and aPTT ≤ 1.5 x ULN.
11. Creatinine clearance > 30 mL/min by Cockcroft-Gault formula.
12. No other active malignancy.
13. For female patients of childbearing potential and male patients with partners of childbearing potential agreement (by patient and/or partner) to use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 6 months after trial completion.
14. Signed informed consent.
15. Ability to comply with the protocol.
16. Systolic ≥80.

Exclusion Criteria:

1. Uncontrolled concomitant disease.
2. History of severe autoimmune disease.
3. Treatment with systemic immunostimulatory agents within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment (with the exception of checkpoint blockade therapy).
4. Treatment with systemic corticosteroids or other systemic immunosuppressive medications within past 4 weeks or 5 half-lives whichever is shorter.
5. Pregnant and/or lactating women.
6. Patients unable to tolerate checkpoint inhibitor therapy.
7. Grade 3 or 4 non-hematological, treatment-related AEs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Beginning of treatment to up to 12 months after beginning of treatment.
  A dose limiting toxicity (DLT) will be defined as a treatment related grade 3-4 non-hematologic toxicity and will require dose de-escalation. If a DLT does not resolve within 5 days, is not responsive to management, or occurs at the lowest dose level (1 million IU IL-2) after de-escalation then that patient will be removed from trial and the therapy will be deemed intolerable. Therapy will be deemed safe and tolerable if no greater than 33% of patients find the treatment intolerable.

SECONDARY OUTCOMES:
Disease free survival | Beginning of treatment to up to 12 months after beginning of treatment.
  Disease free survival will be summarized with Kaplan-Meier plots to describe the outcome of patients treated on this protocol. The median DFS time will be estimated using standard life table methods.

CONTACTS AND LOCATIONS:
Overall Officials: Arta Monjazeb, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No